CLINICAL TRIAL: NCT04828798
Title: Directional Versus Nondirectional Deep Brain Stimulation of the VIM Thalamic Nucleus for Essential Tremor: Assessment of Therapeutic Window, Speech, Gait and Balance
Brief Title: Directional Versus Nondirectional DBS for ET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Matthew Brodsky, Associate Professor of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00020724
Record Dates: First submitted 2021-02-08; First posted 2021-04-02 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: Double-blinded crossover design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Directional deep brain stimulation (Active Comparator): Deep brain stimulation delivered in a directional manner within an axial plane
  Interventions: Device: Deep brain stimulation of the VIM Thalamic nuclei
- Nondirectional deep brain stimulation (Active Comparator): Deep brain stimulation delivered in a nondirectional manner within an axial plane
  Interventions: Device: Deep brain stimulation of the VIM Thalamic nuclei

INTERVENTIONS:
Device: Deep brain stimulation of the VIM Thalamic nuclei — Deep brain stimulation of the thalamus, in a directional and nondirectional manner

SUMMARY:
This will be a single center (OHSU) proof of concept trial to demonstrate that directional deep brain stimulation (DBS) creates a larger therapeutic window for the treatment of essential tremor (ET), effectively treats ET, and minimizes effects on speech, gait and balance compared to nondirectional DBS.

DETAILED DESCRIPTION:
Specific Aims:

1. To compare the therapeutic window (TW) of directional versus nondirectional deep brain stimulation for treatment of tremor.

   Hypothesis: directional DBS will result in a wider TW than nondirectional DBS.
2. To compare the effects of directional versus nondirectional DBS on speech Hypothesis: Objective and subjective speech impairment will occur to a greater extent in nondirectional DBS versus directional DBS optimized for tremor control.
3. To compare the effects of directional versus nondirectional DBS on balance and gait Hypothesis: Objective and subjective balance and gait impairment will occur to a greater extent in nondirectional DBS versus directional DBS optimized for tremor control.
4. To assess efficacy for tremor of nondirectional and directional DBS in an optimized programming configuration Hypothesis: both directional and nondirectional DBS will significantly improve tremor compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* A tremor syndrome of bilateral upper limb action tremor with at least 3 years' duration

Exclusion Criteria:

* Patients who have decided not to receive DBS for control of their medication-refractory essential tremor.
* Patients with secondary tremor (ie not Essential Tremor), such as side effects from medications, secondary to another identified neurologic disease (eg multiple sclerosis, -----Parkinson's disease, dystonia).
* Prior history of deep brain stimulation.
* Prior history of thalamotomy.
* A history or signs of dystonia, ataxia or parkinsonism.
* Task specific tremor.
* Orthostatic tremor.
* Patients with cardiac pacemakers, defibrillators, or neurostimulators.
* Patients who require MRI, ECT, rTMS, or diathermy.
* Subjects with other type of neurological disease or injury.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic window | 3 months
  Range of therapeutic current from clinical improvement to side effect threshold, measured in milliamps, within a range of 0.0 to 5.0 milliamps

SECONDARY OUTCOMES:
Improvement of tremor | 3 months
  Change in The Essential Tremor Rating Scale (TETRAS) combined score. Range = 0 to112. Higher score = worse outcome.
Compare the effects of directional versus nondirectional DBS on self perception of speech | 3 months
  Self Perception of speech: Subjects will rate their "ability to speak" on a VAS (from 0 [normal] to 100 mm [worst]) in each condition.
Compare the effects of directional versus nondirectional DBS on balance and gait | 3 months
  The Activities-specific Balance Confidence (ABC) scale is a 16-item self-report measure in which participants rate their balance confidence on a 0-100 scale (0 = 0 no confidence, 100 = 100 complete confidence).
Compare the effects of directional versus nondirectional DBS on perceptual assessment of voice and speech | 3 months
  Perceptual assessment of voice and speech will be completed with listeners judging a reading sample using a 100mm Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No